CLINICAL TRIAL: NCT01668875
Title: Acute Hemodynamic and Ventilatory Responses to Head-down 30° Postural Drainage Position in Critically Traumatic Patients
Brief Title: Hemodynamic and Ventilatory Responses to Head-down Postural Drainage Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kantharakorn Hongrattana, Principal vinvestigator, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KKU-AMS-PT
Record Dates: First submitted 2012-06-25; First posted 2012-08-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Traumatic Blunt Chest and/or Blunt Abdominal Injury
Keywords: head down postural drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment condition (Experimental): In intervention period patients were received head-down 30 degree postural drainage position for 10 min.
  Interventions: Other: Head down 30 degree postural drainage position
- Sham condition (Experimental): In intervention period patients were received horizontal supine lying for 10 min.
  Interventions: Other: Horizontal supine lying

INTERVENTIONS:
Other: Head down 30 degree postural drainage position — supine head down 30 degree on tilt table (intervention period in the treatment condition)
  Arms: Treatment condition
Other: Horizontal supine lying — horizontal supine lying on tilt table (intervention period in the sham condition)
  Arms: Sham condition

SUMMARY:
The purpose of this study is to explore acute hemodynamic and ventilatory responses to head-down 30 degree postural drainage position in patients with blunt chest and/or abdominal injury in the traumatic intensive care unit.

DETAILED DESCRIPTION:
Study Protocol The study protocol consisted of 2 conditions: treatment condition (A) and sham condition (B). The order of the conditions was randomly assigned to either the treatment or sham for the first round and vise versa in the second round in a balanced cross-over design (A-B-B-A) so there were four sets of measurements per patient.

For the treatment condition (A), the study consists of three consecutive periods 1) baseline period: 10 minutes rest in horizontal supine lying 2) intervention period: 10 minutes rest in head-down 30 degree supine lying 3) recovery period: return to horizontal supine lying and rest for 10 minutes . For the Sham condition (B), the study was performed with a similar procedure except the intervention period consisted of horizontal supine lying.

Hemodynamic and ventilatory parameter were recorded at the start of each period (0 min) and every 2 minute until end of each period for both conditions. Hemodynamic and ventilatory dependent variables were heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), electrocardiography (ECG), central venous pressure (CVP), respiratory rate (RR), oxygen saturation (SpO2), tidal volume (VT), minute ventilation (VE), dynamic lung compliance (Cdyn) and end-tidal expiratory pressure of CO2 (PETCO2). Subjects were rested between each condition. Subjects were suctioned via endotracheal tube to clear airway at 10 minutes before study commencement of either A-B or B-A.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilator dependence
* Stable cardiopulmonary function at rest (HR 60-100 beats/min, systolic BP 90-140 mmHg and diastolic BP 60-90 mmHg and SpO2>95%. RR 10-20 breath/min

Exclusion Criteria:

* Spine disorders such as spine fracture, HNP, spondylolisthesis, whiplash syndrome, stenosis and spondylosis
* Fracture of upper and/or lower limbs
* Underlying acute or chronic cardiopulmonary diseases
* Craniotomy or craniectomy
* Unstable intracranial pressure, ICP>12 cmH2O
* Uncontrolled pain

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change of heart rate (HR) from baseline. | measured every 2 minutes during each phase
  Heart rate (HR) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of systolic blood pressure (SBP) from baseline. | measured every 2 minutes during each phase
  Systolic blood pressure (SBP) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of diastolic blood pressure (DBP) from baseline. | measured every 2 minutes during each phase
  Diastolic blood pressure (DBP) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of mean arterial pressure (MAP) from baseline. | measured every 2 minutes during each phase
  Mean arterial pressure (MAP) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of central venous pressure (CVP) from baseline. | measures every 2 minutes in each phase
  central venous pressure (CVP) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of respiratory rate (RR) from baseline. | measures every 2 minutes in each phase
  respiratory rate (RR) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of tidal volume (VT) from baseline | measured every 2 minutes during each phase
  tidal volume (VT) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of minute ventilation (VE) from baseline | measured every 2 minutes during each phase
  minute ventilation (VE) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of dynamic lung compliance (Cdyn) from baseline. | measured every 2 minutes during each phase
  dynamic lung compliance (Cdyn) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of end-tidal expiratory pressure of carbon dioxide (PETCO2) from baseline | measured every 2 minutes during each phase
  end-tidal expiratory pressure of carbon dioxide (PETCO2) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).
Change of oxygen saturation (SpO2) from baseline | measured every 2 minutes during each phase
  oxygen saturation (SpO2) was recorded 3 times every 2 minute in each phase, each phase will have 10 minutes and each condition will have 3 phases (baseline, intervention, and recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Mr.Kantharakorn Hongrattana, master, Principal Investigator — Department of Physical Therapy, Khon Kaen Hospital
Locations (1):
- Khon Kaen Hospital, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Hongrattana G, Reungjui P, Jones CU. Acute hemodynamic responses to 30 degrees head-down postural drainage in stable, ventilated trauma patients: a randomized crossover trial. Heart Lung. 2014 Sep-Oct;43(5):399-405. doi: 10.1016/j.hrtlng.2014.01.011. Epub 2014 Mar 19. PMID 24655936